CLINICAL TRIAL: NCT02264808
Title: Clinical Utility of Serum Biomarkers for the Management of Neonatal Hypoxic Ischemic Encephalopathy (HIE).
Brief Title: Developmental Outcomes
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201400699
Record Dates: First submitted 2014-10-06; First posted 2014-10-15 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Hypoxic-Ischemic Encephalopathy
MeSH Terms: conditions — Hypoxia-Ischemia, Brain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Biomarkers will be compared to developmental outcomes, however these blood samples were already obtained through IRB#504-2011
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Developmental outcomes: A developmental assessment (Bayley-III) of children 18-20 months who already enrolled in Florida Neonatal Neurologic Network. As part of this previous study, these children were born with Hypoxic Ischemic Encephalopathy (HIE) and underwent therapeutic cooling after birth.
  Interventions: Other: Developmental Outcomes

INTERVENTIONS:
Other: Developmental Outcomes — A Bayley-III developmental assessment will be performed study subjects at age 18-20 months

SUMMARY:
Determine whether the concentrations of UCH-L1 and GFAP measured in umbilical cord blood and in blood 0-6 hours postnatal accurately predict the extent of neurodevelopmental deficits and/or death at 18-20 months.

DETAILED DESCRIPTION:
Children born with Hypoxic Ischemic Encephalopathy (HIE) and already enrolled in IRB #504-2011 will be seen for a developmental follow-up at 18-20 months of age. The developmental assessment tool that will be used is called the Bayley Scales of Infant and Toddler Development: 3rd Edition (Bayley-III) Screening Test. The results of this test will then be compared to the child's HIE biomarkers concentrations already obtained at birth.

ELIGIBILITY:
Inclusion Criteria:

* children already enrolled in IRB#504-2011
* 18-20 months of age

Exclusion Criteria:

* none

Ages: 18 Months to 20 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children 18-20 months of age born with Hypoxic Ischemic Encephalopathy (HIE)
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2018-12-03 (Actual); Study Completion 2018-12-03 (Actual)

PRIMARY OUTCOMES:
Bayley-III developmental assessment in children, with Hypoxic Ischemic Encephalopathy (HIE) diagnosis at birth, at 18-20 months of age | 2 years
  Compare Developmental Outcomes to HIE Biomarker concentrations at birth

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Weiss, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States